CLINICAL TRIAL: NCT05007587
Title: Lenvatinib Combined With Hepatic Arterial Infusion of Modified FOLFOX Regimen Versus Lenvatinib Combined With Hepatic Arterial Infusion of ROX Regimen in the Treatment of Advanced Hepatocellular Carcinoma
Brief Title: Lenvatinib Plus HAIC of Modified FOLFOX Regime vs Lenvatinib Plus HAIC of ROX Regime in Patients With Advanced HCC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Zhejiang Cancer Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Shaoxing People's Hospital (Other); The Third Affiliated Hospital of Wenzhou Medical University (Other); Jinhua Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZJPIRB-2021-211
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2021-08-16 (Actual); Status verified 2021-06

CONDITIONS: Hepatocellular Carcinoma Stage IIIa
Keywords: Lenvatinib; HAIC; HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; folfirinox

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized controlled study
Who Masked: Participant
Masking Description: 60 HCC participants were divided into test group and control group by random drawing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lenvatinib，Then HAIC of mFOLFOX regimen (Experimental): Cohort1：Participants were treated with 8mg lenvatinib (weight<60kg) or 12mg lenvatinib (weight>60kg) orally once daily on days 1 through 21, and HAIC regimen was performed every 3 weeks. The mFOLFOX regimen was administered via hepatic artery: oxaliplatin , 85mg/m2 , from hour 0 to 2 on day1 ; leucovorin , 400mg/m2 , from hour 2 to 3 on day 1 ; fluorouracil , 400mg/m2 , bolus at hour 3 ; and 2400mg/m2 over 46 hours on days 1 and 2.
  Interventions: Drug: Lenvatinib; Drug: mFOLFOX regimen
- Lenvatinib，Then HAIC of ROX regimen (Experimental): Cohort2：Participants were treated with 8mg lenvatinib (weight<60kg) or 12mg lenvatinib (weight>60kg) orally once daily on days 1 through 21, and HAIC regimen was performed every 3 weeks. The ROX regimen was administered via hepatic artery: oxaliplatin , 100mg/m2 , from hour 0 to 4 on day1 ;raltitrexed , 3mg/m2 , from hour 4 to 5 on day 1.
  Interventions: Drug: Lenvatinib; Drug: ROX regimen

INTERVENTIONS:
Drug: Lenvatinib — 8mg lenvatinib (weight<60kg) or 12mg lenvatinib (weight>60kg) QD
  Other Names: LENVIMA
Drug: mFOLFOX regimen — HAIC was performed every 3 weeks. The mFOLFOX regimen was administered via hepatic artery: oxaliplatin , 85mg/m2 , from hour 0 to 2 on day1 ; leucovorin , 400mg/m2 , from hour 2 to 3 on day 1 ; fluorouracil , 400mg/m2 , bolus at hour 3 ; and 2400mg/m2 over 46 hours on days 1 and 2.3mg/m2 , from hour 4 to 5 on day 1.
  Other Names: Oxaliplatin+Leucovorin+Fluorouracil
  Arms: Lenvatinib，Then HAIC of mFOLFOX regimen
Drug: ROX regimen — HAIC was performed every 3 weeks. The ROX regimen was administered via hepatic artery: oxaliplatin , 100mg/m2 , from hour 0 to 4 on day1 ;raltitrexed , 3mg/m2 , from hour 4 to 5 on day 1.
  Other Names: Raltitrexed+Oxaliplatin
  Arms: Lenvatinib，Then HAIC of ROX regimen

SUMMARY:
Lenvatinib Plus Hepatic Arterial Infusion of Modified FOLFOX Regime vs Lenvatinib Plus Hepatic Arterial Infusion of Oxaliplatin Plus Raltitrexed in Patients with Advanced Hepatocellular Carcinoma

DETAILED DESCRIPTION:
Hepatic arterial infusion chemotherapy is one of the important means for the treatment of advanced liver cancer. A multicenter randomized controlled study has confirmed that modified FOLFOX hepatic arterial infusion chemotherapy can significantly improve the prognosis of patients with advanced liver cancer and prolong the survival period of patients. The 2020 edition of CSCO guidelines for the diagnosis and treatment of liver cancer has recommended oxaliplatin based FOLFOX arterial infusion regimen as the first-line treatment of advanced liver cancer. FOLFOX regimen is safe and effective, but fluorouracil needs more than 46 hours of long-term infusion, patients have difficulty in moving during catheterization, and increase the risk of thrombosis, so it is urgent to find a short-term infusion of fluorouracil. As a new antimetabolic drug, raltitrexed can be used for short-term infusion, and its plasma concentration half-life is longer than that of fluorouracil. Previous studies have shown that compared with FOLFOX arterial infusion regimen, oxaliplatin combined with raltitrexed regimen has longer overall survival (OS) and progression free survival (PFS) in the treatment of advanced liver cancer. In addition, as an advanced liver cancer, lenvastinib has been recommended as a targeted drug for the first-line treatment of advanced HCC. This study intends to explore the efficacy and safety of modified FOLFOX regimen compared with oxaliplatin combined with raltitrexed (Rox regimen) in the treatment of lenvastinib combined with HAIC, so as to provide more clinical schemes for further improving the survival rate of patients with advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary participation and informed consent, aged 18-75;
2. Patients with HCC confirmed by histopathology or meeting the clinical diagnostic criteria in the 2019 edition of the diagnostic and therapeutic criteria for primary liver cancer;
3. BCLC stage C patients with vascular invasion and without extrahepatic metastasis;
4. Child Pugh liver function classification: A or B grade;
5. ECOG physical strength score was 0-2 points;
6. No previous systemic or local treatment, and the expected survival time is more than 3 months;
7. According to recist1.1, the patient must have at least one measurable target lesion that has passed CT or MRI examination, and the tumor imaging evaluation was conducted within 2 weeks before receiving the study drug;
8. Full organ and bone marrow function: WBC ≥ 3.0 × 109/L； NE≥1.5 × 109/L； PLT≥75 × 109/L； Liver and kidney function ALT and AST ≤ 5uln; TBIL≤2ULN； Albumin ≥ 28g / L; Cr≤1.5 ULN； International normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) exceeding the normal control range ≤ 4 seconds;

Exclusion Criteria:

1. Hepatocholangiocarcinoma, mixed cell carcinoma and fibrolamellar cell carcinoma are known;
2. Uncontrollable ascites, hepatic encephalopathy or esophageal variceal bleeding;
3. Patients with hypertension who can not be reduced to normal range after antihypertensive drug treatment (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
4. Patients with myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia, myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmia (QTc interval ≥ 450 ms) (QTc interval was calculated by fridericia formula);
5. Patients with history of gastrointestinal bleeding or definite tendency of gastrointestinal bleeding in the past 3 months, such as esophageal varices with bleeding risk, local active ulcer lesions, fecal occult blood ≥ +, can not be included in the group;
6. Pregnant or lactating women, patients with fertility are unwilling or unable to take effective contraceptive measures;
7. patients with a history of HIV infection;
8. The researcher judges other situations that may affect the clinical research and the judgment of research results;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate and Disease Control Rate of the HCC Participants | from admission to discharge, up to 4 weeks
  ORR and DCR are validated indicators of the short-term clinical effects of hepatocellular carcinoma

SECONDARY OUTCOMES:
Overall Survival and Progression-free Survival of the HCC Participants | six months and twelve months
  OS and PFS are validated indicators of the long-term clinical effects of hepatocellular carcinoma
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | from admission to discharge, up to 4 weeks
  Treatment-Related Adverse Events are important indicators of the safety for tumor treatment

OTHER OUTCOMES:
Weight and Height | from admission to discharge, up to 1 week
  Weight and Height will be combined to report BMI in kg/m^2
Age | from admission to discharge, up to 1 week
  Age is divided into >50 and ≤50
Sex | from admission to discharge, up to 1 week
  Sex is divided into Male and Female
ECOG score | from admission to discharge, up to 1 week
  ECOG score is divided into 0,1,2
Tumor size | from admission to discharge, up to 1 week
  Tumor size is divided into >10cm and ≤10cm
Tumor number | from admission to discharge, up to 1 week
  Tumor number is divided into single and multiple
AFP | from admission to discharge, up to 1 week
  AFP is divided into >1000ug/L and ≤1000ug/L
Portal vein invasion | from admission to discharge, up to 1 week
  Portal vein invasion is divided into Vp1-2, Vp3, Vp4
Extrahepatic spread | from admission to discharge, up to 1 week
  Extrahepatic spread is divided into Yes and No
Hepatitis B infection | from admission to discharge, up to 1 week
  Hepatitis B infection is divided into Yes and No

CONTACTS AND LOCATIONS:
Overall Officials: Jiaping Zheng, Doctor, Study Chair — Zhejiang Cancer Hospital
Locations (1):
- The Cancer Hospital of the University of Chinese Academy of Sciences（Zhejiang Cancer Hospital）, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Result] Global Burden of Disease Cancer Collaboration; Fitzmaurice C, Allen C, Barber RM, Barregard L, Bhutta ZA, Brenner H, Dicker DJ, Chimed-Orchir O, Dandona R, Dandona L, Fleming T, Forouzanfar MH, Hancock J, Hay RJ, Hunter-Merrill R, Huynh C, Hosgood HD, Johnson CO, Jonas JB, Khubchandani J, Kumar GA, Kutz M, Lan Q, Larson HJ, Liang X, Lim SS, Lopez AD, MacIntyre MF, Marczak L, Marquez N, Mokdad AH, Pinho C, Pourmalek F, Salomon JA, Sanabria JR, Sandar L, Sartorius B, Schwartz SM, Shackelford KA, Shibuya K, Stanaway J, Steiner C, Sun J, Takahashi K, Vollset SE, Vos T, Wagner JA, Wang H, Westerman R, Zeeb H, Zoeckler L, Abd-Allah F, Ahmed MB, Alabed S, Alam NK, Aldhahri SF, Alem G, Alemayohu MA, Ali R, Al-Raddadi R, Amare A, Amoako Y, Artaman A, Asayesh H, Atnafu N, Awasthi A, Saleem HB, Barac A, Bedi N, Bensenor I, Berhane A, Bernabe E, Betsu B, Binagwaho A, Boneya D, Campos-Nonato I, Castaneda-Orjuela C, Catala-Lopez F, Chiang P, Chibueze C, Chitheer A, Choi JY, Cowie B, Damtew S, das Neves J, Dey S, Dharmaratne S, Dhillon P, Ding E, Driscoll T, Ekwueme D, Endries AY, Farvid M, Farzadfar F, Fernandes J, Fischer F, G/Hiwot TT, Gebru A, Gopalani S, Hailu A, Horino M, Horita N, Husseini A, Huybrechts I, Inoue M, Islami F, Jakovljevic M, James S, Javanbakht M, Jee SH, Kasaeian A, Kedir MS, Khader YS, Khang YH, Kim D, Leigh J, Linn S, Lunevicius R, El Razek HMA, Malekzadeh R, Malta DC, Marcenes W, Markos D, Melaku YA, Meles KG, Mendoza W, Mengiste DT, Meretoja TJ, Miller TR, Mohammad KA, Mohammadi A, Mohammed S, Moradi-Lakeh M, Nagel G, Nand D, Le Nguyen Q, Nolte S, Ogbo FA, Oladimeji KE, Oren E, Pa M, Park EK, Pereira DM, Plass D, Qorbani M, Radfar A, Rafay A, Rahman M, Rana SM, Soreide K, Satpathy M, Sawhney M, Sepanlou SG, Shaikh MA, She J, Shiue I, Shore HR, Shrime MG, So S, Soneji S, Stathopoulou V, Stroumpoulis K, Sufiyan MB, Sykes BL, Tabares-Seisdedos R, Tadese F, Tedla BA, Tessema GA, Thakur JS, Tran BX, Ukwaja KN, Uzochukwu BSC, Vlassov VV, Weiderpass E, Wubshet Terefe M, Yebyo HG, Yimam HH, Yonemoto N, Younis MZ, Yu C, Zaidi Z, Zaki MES, Zenebe ZM, Murray CJL, Naghavi M. Global, Regional, and National Cancer Incidence, Mortality, Years of Life Lost, Years Lived With Disability, and Disability-Adjusted Life-years for 32 Cancer Groups, 1990 to 2015: A Systematic Analysis for the Global Burden of Disease Study. JAMA Oncol. 2017 Apr 1;3(4):524-548. doi: 10.1001/jamaoncol.2016.5688. PMID 27918777
- [Result] Cheng AL, Kang YK, Chen Z, Tsao CJ, Qin S, Kim JS, Luo R, Feng J, Ye S, Yang TS, Xu J, Sun Y, Liang H, Liu J, Wang J, Tak WY, Pan H, Burock K, Zou J, Voliotis D, Guan Z. Efficacy and safety of sorafenib in patients in the Asia-Pacific region with advanced hepatocellular carcinoma: a phase III randomised, double-blind, placebo-controlled trial. Lancet Oncol. 2009 Jan;10(1):25-34. doi: 10.1016/S1470-2045(08)70285-7. Epub 2008 Dec 16. PMID 19095497
- [Result] Benson AB, D'Angelica MI, Abbott DE, Abrams TA, Alberts SR, Anaya DA, Anders R, Are C, Brown D, Chang DT, Cloyd J, Covey AM, Hawkins W, Iyer R, Jacob R, Karachristos A, Kelley RK, Kim R, Palta M, Park JO, Sahai V, Schefter T, Sicklick JK, Singh G, Sohal D, Stein S, Tian GG, Vauthey JN, Venook AP, Hammond LJ, Darlow SD. Guidelines Insights: Hepatobiliary Cancers, Version 2.2019. J Natl Compr Canc Netw. 2019 Apr 1;17(4):302-310. doi: 10.6004/jnccn.2019.0019. PMID 30959462
- [Result] Spallanzani A, Orsi G, Andrikou K, Gelsomino F, Rimini M, Riggi L, Cascinu S. Lenvatinib as a therapy for unresectable hepatocellular carcinoma. Expert Rev Anticancer Ther. 2018 Nov;18(11):1069-1076. doi: 10.1080/14737140.2018.1524297. Epub 2018 Sep 21. PMID 30220234
- [Result] Song DS, Song MJ, Bae SH, Chung WJ, Jang JY, Kim YS, Lee SH, Park JY, Yim HJ, Cho SB, Park SY, Yang JM. A comparative study between sorafenib and hepatic arterial infusion chemotherapy for advanced hepatocellular carcinoma with portal vein tumor thrombosis. J Gastroenterol. 2015 Apr;50(4):445-54. doi: 10.1007/s00535-014-0978-3. Epub 2014 Jul 16. PMID 25027973
- [Result] Obi S, Sato S, Kawai T. Current Status of Hepatic Arterial Infusion Chemotherapy. Liver Cancer. 2015 Sep;4(3):188-99. doi: 10.1159/000367746. Epub 2015 Aug 12. PMID 26674592
- [Result] Lyu N, Kong Y, Mu L, Lin Y, Li J, Liu Y, Zhang Z, Zheng L, Deng H, Li S, Xie Q, Guo R, Shi M, Xu L, Cai X, Wu P, Zhao M. Hepatic arterial infusion of oxaliplatin plus fluorouracil/leucovorin vs. sorafenib for advanced hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):60-69. doi: 10.1016/j.jhep.2018.02.008. Epub 2018 Feb 20. PMID 29471013
- [Result] Zhuang BW, Li W, Xie XH, Hu HT, Lu MD, Xie XY. Sorafenib versus hepatic arterial infusion chemotherapy for advanced hepatocellular carcinoma: a systematic review and meta-analysis. Jpn J Clin Oncol. 2019 Sep 1;49(9):845-855. doi: 10.1093/jjco/hyz069. PMID 31063184
- [Result] Chen S, Zhang K, Liu W, Yu W. Hepatic arterial infusion of oxaliplatin plus raltitrexed in patients with intermediate and advanced stage hepatocellular carcinoma: A phase II, single-arm, prospective study. Eur J Cancer. 2020 Jul;134:90-98. doi: 10.1016/j.ejca.2020.03.032. Epub 2020 Jun 1. PMID 32497895
- [Result] He M, Li Q, Zou R, Shen J, Fang W, Tan G, Zhou Y, Wu X, Xu L, Wei W, Le Y, Zhou Z, Zhao M, Guo Y, Guo R, Chen M, Shi M. Sorafenib Plus Hepatic Arterial Infusion of Oxaliplatin, Fluorouracil, and Leucovorin vs Sorafenib Alone for Hepatocellular Carcinoma With Portal Vein Invasion: A Randomized Clinical Trial. JAMA Oncol. 2019 Jul 1;5(7):953-960. doi: 10.1001/jamaoncol.2019.0250. PMID 31070690